CLINICAL TRIAL: NCT00483496
Title: Evaluation of the Protection Activity of Microfine Ti02, Pigmentary Ti02 and Bisoctrizole and Their Combinations in Voluntary Patients With SU: Phase II Photoprovocation Test
Brief Title: Evaluation of the Protection Activity of Microfine Titanium Dioxide (Ti02), Pigmentary Ti02 and Bisoctrizole and Their Combinations in Voluntary Patients With Idiopathic Solar Urticaria (SU)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orfagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: V00096 CR 205 (ORF)
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Idiopathic Solar Urticaria
MeSH Terms: interventions — titanium dioxide; Single Person

STUDY DESIGN:
Who Masked: Investigator

ARMS (1):
- V0096CR actives and vehicle (Experimental): Each patient received each one of the 8 test products on their respective randomly allocated sites on grid (grid to be applied on the back skin; 1 product by grid window).
  Single application of the test materials at the dosage of 2mg/cm² (total of 8 treated sites), prior to irradiation using a solar simulator.
  Interventions: Drug: Titanium dioxide (Ti02) microfine 12.15% alone (formula RV3131A-MV1209); Drug: Ti02 pigmentary 3% alone (formula RV3131A-MV1211); Drug: bisoctrizole 10% alone (formula RV3131A-MV1237); Drug: Ti02 microfine 12.15% + Ti02 pigmentary 3% (formula RV3131A-MV1213); Drug: Ti02 microfine 12.15% + bisoctrizole 10% (formula RV3131A-MV1329); Drug: Ti02 pigmentary 3% + bisoctrizole 10% (formula RV3131A-MV1212); Drug: Ti02 microfine 12.15% + Ti02 pigmentary 3% + bisoctrizole 10% [V0096 CR (formula RV3131A-MV1166)]; Drug: V0096 CR vehicle (formula RV3131A-MV1197)

INTERVENTIONS:
Drug: Titanium dioxide (Ti02) microfine 12.15% alone (formula RV3131A-MV1209)
Drug: Ti02 pigmentary 3% alone (formula RV3131A-MV1211)
Drug: bisoctrizole 10% alone (formula RV3131A-MV1237)
Drug: Ti02 microfine 12.15% + Ti02 pigmentary 3% (formula RV3131A-MV1213)
Drug: Ti02 microfine 12.15% + bisoctrizole 10% (formula RV3131A-MV1329)
Drug: Ti02 pigmentary 3% + bisoctrizole 10% (formula RV3131A-MV1212)
Drug: Ti02 microfine 12.15% + Ti02 pigmentary 3% + bisoctrizole 10% [V0096 CR (formula RV3131A-MV1166)]
Drug: V0096 CR vehicle (formula RV3131A-MV1197)

SUMMARY:
Commercially available external photoprotectors (EP) do not provide adequate protection against ultraviolet A (UVA) and visible wavelengths. The proposed medicinal product V0096 CR (formula RV3131A-MV1166) is a broad spectrum EP (bsEP). The rationale for the use of V0096 CR (formula RV3131A-MV1166) in the proposed condition is based on its ability to broadly block the UVA radiations and visible light that are known to trigger solar urticaria (SU).

ELIGIBILITY:
Inclusion Criteria:

* Male or female voluntary patients at least 18 years old
* For female patients with child-bearing potential, negative pregnancy test at baseline
* Patients with a clinical and photobiological diagnosis of idiopathic SU
* Patients with no underlying condition, or with underlying conditions provided that these conditions are stable and under control
* Patients able to follow instructions
* Written informed consent from the patients

Exclusion Criteria:

* Children (less than 18 years old)
* Pregnant or lactating women
* Women with a positive pregnancy test at baseline
* Patients with spontaneous occurrence of SU lesions on the back within 3 days prior to study entry
* Patients with a known allergy to one of the ingredients contained in the test products
* Patients who have applied EP to back skin over the previous 2 weeks before study entry
* Patients who have applied topical corticosteroids to back skin within 7 days prior to study entry
* Patients who have applied an emollient including white soft paraffin on back skin within 2 days prior to study entry
* Patients with systemic exposure to corticosteroids, anti-inflammatories or other immunosuppressive agents within the last 4 weeks prior to study entry
* Patients with oral antihistamines within the last 2 days prior to study entry
* Patients who have been administered systemic or topical photoactive medications for phototherapy or phototherapy alone within 1 week prior to study entry
* Patients with an unstable or non-controlled underlying condition
* Patients who are not able to follow instructions
* Patients who have participated in a study within the 3 months prior to study entry
* Patients who refuse to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Dupuy, Dr, Study Director — Orfagen; James Ferguson, Pr, Principal Investigator — Ninewells Hospital
Locations (3):
- United States (2):
  - Henry Ford Medical Center, Detroit, Michigan
  - St Luke's Roosevelt Hospital Center, New York, New York
- Ninewells Hospital, Dundee, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Each patient received the 8 test products on the 8 test areas of the randomly allocated grid.
Period: Overall Study
Arm/Group | Experimental
Started | 16
Completed | 15
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 50.2 [26 to 82]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 10
  United Kingdom | 5

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Minimal Urticaria Dose (MUD) on Each Test Site, After Application of the Test Products
Description: MUD was defined as the minimal dose for occurrence of objective signs of SU (wheal, flare) under exposure to the solar simulator. Results are expressed as photodermatosis protection factor (PPF), calculated by dividing the MUD of protected skin (sessions 2 to 5) by the MUD of the unprotected skin (session 1) in each treatment group.
  Procedure: At baseline, 4 grids of 8 adjacent test areas on the patient back were defined. The defined test areas of each grid were applied with the respective test products by the investigating staff at the beginning of each session, according to a predefined randomisation schedule. Grids were sequentially irradiated one by one with 1 MUD (session 2) , 3 MUD (session 3) , 5 MUD (session 4), and 7 MUD (session 5), respectively. After product removal at each session, patients were observed for 30 min for the development of SU lesions. Final reading of all areas was performed at the end of each session, by the investigator masked to product site assignment.
Time Frame: During each one of the 5 sessions, at study day
Measure: Mean (Full Range); unit: Photodermatosis Protection Factor
Groups:
- V0096; Ti02Pig + Bisoctrizole; TiO2 Micro + Bisoctrizole; TiO2Pig + TiO2Micro; Bisoctrizole; TiO2 Micro; TiO2Pig; Vehicle: Each patient received each one of the 8 test products on their respective randomly allocated sites on grid (grid to be applied on the back skin; 1 product by grid window).
Arm/Group | V0096 | Ti02Pig + Bisoctrizole | TiO2 Micro + Bisoctrizole | TiO2Pig + TiO2Micro | Bisoctrizole | TiO2 Micro | TiO2Pig | Vehicle
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15
Photodermatosis Protection Factor | 4.33 [1.00 to 9.00] | 3.93 [1.00 to 9.00] | 3.80 [1.00 to 9.00] | 3.67 [1.00 to 9.00] | 3.53 [1.00 to 9.00] | 3.27 [1.00 to 9.00] | 2.33 [1.00 to 7.00] | 1.93 [1.00 to 3.00]

2. Secondary Outcome: Adverse Events
Time Frame: through study completion
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 15
Participants | 1

ADVERSE EVENTS:
Arm/Group | Experimental
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=15)
URTICARIA HEAT (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications relating to the TRIAL and results therefrom are subject to prior mutual agreement of the SPONSOR and the INVESTIGATOR.